CLINICAL TRIAL: NCT02818114
Title: Peer Enhanced Exposure Therapy (PEET)
Brief Title: Peer Enhanced Prolonged Exposure
Acronym: PEET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2188-P
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: PTSD
Keywords: PTSD; Prolonged Exposure; Peer Support
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Peer specialist led individual education and support for veterans receiving Prolonged Exposure Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PEET (Experimental): Peer support interventions as an adjunct to prolonged exposure
  Interventions: Behavioral: Peer Enhanced Prolonged Exposure

INTERVENTIONS:
Behavioral: Peer Enhanced Prolonged Exposure — Peer support interventions as adjunct to prolonged exposure
  Other Names: PEET

SUMMARY:
The investigators plan to develop and test an intervention using peer specialists (Veterans who have managed PTSD and completed PE) to provide support services for Veterans using prolonged exposure therapy.

DETAILED DESCRIPTION:
The investigators will use qualitative data from Veterans and PE providers to revise the investigators' manualized intervention for peer support services, then complete a feasibility trial to assess the feasibility and acceptability of Peer Enhanced Prolonged Exposure

ELIGIBILITY:
Inclusion Criteria:

* Veteran participants will be individuals appropriate for PE, i.e., :

  * Veterans who are currently seeking PE
  * meet DSM-5 criteria for PTSD or subthreshold PTSD
  * are competent to consent to research

Exclusion Criteria:

* Veteran participants do not have levels of other types of psychopathology that would prevent successful participation in the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10-16 (Actual); Primary Completion 2018-06-16 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette I. Harris, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited from veterans screening for Prolonged Exposure (PE) at a Midwestern VA between 6/2017 and 3/2018. Note that the study was open between 10/2016 and 3/2018, because between 10/2016 and 2/2017 we were enrolling focus groups to refine the intervention to be tested in the clinical trial; the focus groups were not the clinical trial..
Pre-assignment Details: 31 participants were referred by outpatient therapists. 9 were not interested, and 6 did not meet institutional criteria to start PE. 16 consented to interview screening. 5 did not meet criteria to start PE, 2 were lost to follow-up before starting, and one chose not to start PE.
Groups:
- Peer Enhanced Exposure Therapy (PEET): Single Arm Feasibility Trial: Peer Enhanced Prolonged Exposure: Peer support interventions as adjunct to Prolonged Exposure
Period: Overall Study
Arm/Group | Peer Enhanced Exposure Therapy (PEET)
Started | 8
Completed | 7
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- PEET: Single Arm Feasibility Trial: Peer Enhanced Prolonged Exposure: Peer support interventions as adjunct to prolonged exposure
Arm/Group | PEET
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.25 (14.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8
Posttraumatic Stress Disorder Checklist-5 [Mean (Standard Deviation); unit: units on a scale] — Score range is 0-80, with higher scores indicating more PTSD symptoms
  units on a scale | 62.00 (9.70)

OUTCOME MEASURES:

1. Primary Outcome: PE Sessions Attended
Description: Number of PE Sessions attended during 10 weeks of participation in study. 10 is the maximum, 0 is the minimum. Higher numbers of sessions attended are an indication of better engagement in treatment.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: number of PE sessions attended
Groups:
- Peer Enhanced Prolonged Exposure: Standard Prolonged Exposure therapy supplemented by weekly, manualized peer support sessions.
Arm/Group | Peer Enhanced Prolonged Exposure
Number analyzed (Participants) | 8
number of PE sessions attended | 8.63 (2.62)

2. Primary Outcome: Posttraumatic Stress Disorder (PTSD) Checklist-5
Description: Self-report measure of PTSD symptoms; score range is 0-80, with higher scores indicating more PTSD symptoms.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PEET
Number analyzed (Participants) | 8
score on a scale | 33.14 (11.63)
Statistical Analysis 1: Comparison: PEET; This is a single-arm feasibility study. With N=8, formal hypothesis testing is not possible. We were assessing the extent to which veterans would be willing to engage in the intervention, and if the direction of change in symptoms is still in the expected direction when peer support services are added. Outcomes are reported more qualitatively; Test type: Other — Assessment of number of PE sessions attended, review of direction of change in PTSD Checklist scores; As a feasibility trial, tests of statistical significance are not appropriate

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | PEET
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT02818114/Prot_SAP_000.pdf